CLINICAL TRIAL: NCT04570371
Title: Non-Pharmacological Options in Postoperative Hospital-based and Rehabilitation Pain Management: The NOHARM Trial
Brief Title: Non-pharmacological Pain Management After Surgery
Acronym: NOHARM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Andrea Cheville, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-004839; UG3AG067593 (NIH)
Record Dates: First submitted 2020-09-28; First posted 2020-09-30 (Actual); Results first posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Surgical Procedure, Unspecified

STUDY DESIGN:
Intervention Model Description: This is a stepped wedge cluster randomized pragmatic clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Per a stepped-wedge cluster randomized pragmatic clinical trial design, all patients within whole surgical practices will be randomized to implementation tranches in which the intervention will be implemented per the study schedule.
  Interventions: Behavioral: Conversation Guide + Clinical Support
- Control Arm (No Intervention): Per a stepped-wedge cluster randomized pragmatic clinical trial design, all patients within whole surgical practices will be randomized to implementation tranches. The control arm consists of all patients receiving surgery in implementation tranches in which the intervention has not been implemented yet (per the study schedule).

INTERVENTIONS:
Behavioral: Conversation Guide + Clinical Support — The intervention is a bundled intervention (conversation guide + clinician decision support tools) which promotes the solicitation and use of patient preferences for post-surgical, non-pharmacological pain management strategies.
  Arms: Intervention

SUMMARY:
The purpose of this study is to test the impact of a bundled NOHARM Conversation Guide with clinical decision support intervention embedded within an Electronic Health Record (EHR) on pain and function 3 months following surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years of age and older.
* Must be undergoing qualifying surgeries at participating sites.
* Patients under 18 years of age.

Exclusion Criteria:

- Patients under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81938 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Cheville, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Redmond S; Mayo Clinic NOHARM Research Team; Tilburt J, Cheville A. Non-pharmacological Options in Postoperative Hospital-Based and Rehabilitation Pain Management (NOHARM): Protocol for a Stepped-Wedge Cluster-Randomized Pragmatic Clinical Trial. Pain Ther. 2022 Sep;11(3):1037-1053. doi: 10.1007/s40122-022-00393-x. Epub 2022 Jun 3. PMID 35657564

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 13,796 participants were excluded from the study prior to randomization and data collection due to principal investigator discretion.
Units Other Than Participants: Surgical departments
Groups:
- Sequence 1: Per a stepped-wedge cluster randomized pragmatic clinical trial design, all patients within whole surgical practices will be randomized to implementation tranches in which the intervention will be implemented per the study schedule.
  Sequence 1 went live with the intervention during Step 2: Surgical practices offered 4 months of usual care followed by 36 months of intervention. However, patients did not transition from usual care to intervention.
- Sequence 2: Per a stepped-wedge cluster randomized pragmatic clinical trial design, all patients within whole surgical practices will be randomized to implementation tranches in which the intervention will be implemented per the study schedule.
  Sequence 2 went live with the intervention during Step 3. Surgical practices offered 11 months of usual care followed by 29 months of intervention. However, patients did not transition between usual care and intervention.
- Sequence 3: Per a stepped-wedge cluster randomized pragmatic clinical trial design, all patients within whole surgical practices will be randomized to implementation tranches in which the intervention will be implemented per the study schedule.
  Sequence 3 went live with the intervention during Step 4. Surgical practices offered 18 months of usual care followed by 22 months of intervention. However, patients did not transition from usual care to intervention.
- Sequence 4: Per a stepped-wedge cluster randomized pragmatic clinical trial design, all patients within whole surgical practices will be randomized to implementation tranches in which the intervention will be implemented per the study schedule.
  Sequence 4 went live with the intervention during Step 5. Surgical practices offered 25 months of usual care followed by 15 months of intervention. However, patients did not transition from usual care to intervention.
- Sequence 5: Per a stepped-wedge cluster randomized pragmatic clinical trial design, all patients within whole surgical practices will be randomized to implementation tranches in which the intervention will be implemented per the study schedule.
  Sequence 5 went live with the intervention during Step 6. Surgical practices offered 32 months of usual care followed by 8 months of intervention. However, patients did not transition from usual care to intervention.
Period: Step 1: Oct 16 2020 - Feb 28 2021
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5
Started | 1899; 5 Surgical departments | 2378; 5 Surgical departments | 1265; 4 Surgical departments | 721; 4 Surgical departments | 840; 4 Surgical departments
Completed | 1899; 5 Surgical departments | 2378; 5 Surgical departments | 1265; 4 Surgical departments | 721; 4 Surgical departments | 840; 4 Surgical departments
Not Completed | 0; 0 Surgical departments | 0; 0 Surgical departments | 0; 0 Surgical departments | 0; 0 Surgical departments | 0; 0 Surgical departments
Period: Step 2: Mar 1 2021 - Sep 30 2021
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5
Started | 3228; 5 Surgical departments | 3854; 5 Surgical departments | 2112; 4 Surgical departments | 1147; 4 Surgical departments | 1726; 4 Surgical departments
Completed | 3228; 5 Surgical departments | 3854; 5 Surgical departments | 2112; 4 Surgical departments | 1147; 4 Surgical departments | 1726; 4 Surgical departments
Not Completed | 0; 0 Surgical departments | 0; 0 Surgical departments | 0; 0 Surgical departments | 0; 0 Surgical departments | 0; 0 Surgical departments
Period: Step 3: Oct 1 2021 - Apr 30 2022
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5
Started | 3130; 5 Surgical departments | 3660; 5 Surgical departments | 1902; 4 Surgical departments | 1157; 4 Surgical departments | 1500; 4 Surgical departments
Completed | 3130; 5 Surgical departments | 3660; 5 Surgical departments | 1902; 4 Surgical departments | 1157; 4 Surgical departments | 1500; 4 Surgical departments
Not Completed | 0; 0 Surgical departments | 0; 0 Surgical departments | 0; 0 Surgical departments | 0; 0 Surgical departments | 0; 0 Surgical departments
Period: Step 4: May 1 2022 - Nov 30 2022
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5
Started | 3394; 5 Surgical departments | 4038; 5 Surgical departments | 2035; 4 Surgical departments | 1145; 4 Surgical departments | 1715; 4 Surgical departments
Completed | 3394; 5 Surgical departments | 4038; 5 Surgical departments | 2035; 4 Surgical departments | 1145; 4 Surgical departments | 1715; 4 Surgical departments
Not Completed | 0; 0 Surgical departments | 0; 0 Surgical departments | 0; 0 Surgical departments | 0; 0 Surgical departments | 0; 0 Surgical departments
Period: Step 5: Dec 1 2022 - Jun 30 2023
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5
Started | 3486; 5 Surgical departments | 4328; 5 Surgical departments | 2054; 4 Surgical departments | 1233; 4 Surgical departments | 1715; 4 Surgical departments
Completed | 3486; 5 Surgical departments | 4328; 5 Surgical departments | 2054; 4 Surgical departments | 1233; 4 Surgical departments | 1715; 4 Surgical departments
Not Completed | 0; 0 Surgical departments | 0; 0 Surgical departments | 0; 0 Surgical departments | 0; 0 Surgical departments | 0; 0 Surgical departments
Period: Step 6: Jul 1 2023 - Jan 31 2024
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5
Started | 3526; 5 Surgical departments | 4131; 5 Surgical departments | 2017; 4 Surgical departments | 1171; 4 Surgical departments | 1635; 4 Surgical departments
Completed | 3526; 5 Surgical departments | 4131; 5 Surgical departments | 2017; 4 Surgical departments | 1171; 4 Surgical departments | 1635; 4 Surgical departments
Not Completed | 0; 0 Surgical departments | 0; 0 Surgical departments | 0; 0 Surgical departments | 0; 0 Surgical departments | 0; 0 Surgical departments

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Intervention | Total
Number analyzed (Participants) | 25088 | 43054 | 68142
Age, Customized [Count of Participants; unit: Participants]
  Age (category): <=40 | 3681 | 7695 | 11376
  Age (category): 41-50 | 2878 | 4464 | 7342
  Age (category): 51-60 | 4507 | 7039 | 11546
  Age (category): 61-70 | 7236 | 12052 | 19288
  Age (category): 71-80 | 5271 | 9302 | 14573
  Age (category): 80+ | 1515 | 2502 | 4017
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There were two participants in the study who did not provide their gender as male/female.
  Participants
    number analyzed (Participants) | 25087 | 43053 | 68140
    Female | 10429 | 16819 | 27248
    Male | 14658 | 26234 | 40892
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 990 | 1505 | 2495
  Not Hispanic or Latino | 24024 | 41340 | 65364
  Unknown or Not Reported | 74 | 209 | 283
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 185 | 314 | 499
  Asian | 547 | 1009 | 1556
  Native Hawaiian or Other Pacific Islander | 30 | 62 | 92
  Black or African American | 1044 | 1652 | 2696
  White | 22682 | 38971 | 61653
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 600 | 1046 | 1646
Region of Enrollment [Number; unit: participants]
  United States | 25088 | 43054 | 68142
Employment [Count of Participants; unit: Participants]
  Employed | 11229 | 20549 | 31778
  Retired | 10310 | 16528 | 26838
  Not Employed or Student or Military duty | 2341 | 4294 | 6635
  Disabled | 1189 | 1573 | 2762
  Unknown or Not Reported | 19 | 110 | 129
Marital status [Count of Participants; unit: Participants]
  Married | 17015 | 29673 | 46688
  Single | 3772 | 6449 | 10221
  Divorced | 1936 | 3263 | 5199
  Widowed | 1891 | 2825 | 4716
  Life Partnership | 245 | 458 | 703
  Separated | 163 | 247 | 410
  Unknown | 66 | 139 | 205
Education [Count of Participants; unit: Participants]
  Less than high school | 4590 | 7143 | 11733
  High school graduate | 737 | 1230 | 1967
  Some college, vocational school, or associate degree | 7365 | 11660 | 19025
  Bachelor's degree | 5786 | 9175 | 14961
  Master's or Doctoral degree | 4356 | 7068 | 11424
  Unknown | 2254 | 6778 | 9032
Rurality (RUCA code) [Count of Participants; unit: Participants]
  Urban (RUCA 1-3) | 18150 | 29743 | 47893
  Micropolitan (RUCA 4-6) | 2661 | 5297 | 7958
  Small town (RUCA 7-9) | 2284 | 4217 | 6501
  Rural (RUCA 10) | 1835 | 3555 | 5390
  Unknown | 158 | 242 | 400

OUTCOME MEASURES:

1. Primary Outcome: PROMIS-CAT Pain
Description: Change in patient reported pain; measured on scale of 1-100. A higher score indicates a worse outcome.
Time Frame: Baseline (before hospital discharge), 1-,2-, and 3-Months Post-Surgery
Population: Number of participants who answered at least 1 pain followup survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Arm | Intervention
Number analyzed (Participants) | 16819 | 30349
score on a scale
  Baseline | 59.32 (9.92) | 59.96 (9.68)
  Month 1 | 56.94 (9.10) | 56.06 (8.97)
  Month 2 | 53.08 (9.42) | 53.29 (9.39)
  Month 3 | 52.14 (9.43) | 52.43 (9.45)

2. Primary Outcome: PROMIS-CAT Physical Function
Description: Change in patient reported Physical Function; measured on scale of 1-100. A higher score indicates a better outcome.
Time Frame: Baseline (before hospital discharge), 1-,2-, and 3-Months Post-Surgery
Population: Number of participants who answered at least one physical function followup survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Arm | Intervention
Number analyzed (Participants) | 16543 | 29973
score on a scale
  Baseline | 40.50 (9.04) | 39.50 (8.54)
  Month 1 | 38.44 (9.06) | 39.68 (9.19)
  Month 2 | 42.44 (9.75) | 40.79 (10.26)
  Month 3 | 43.84 (9.74) | 41.85 (10.41)

3. Primary Outcome: PROMIS-CAT Anxiety
Description: Change in patient reported Anxiety; measured on scale of 1-100. A higher score indicates a worse outcome.
Time Frame: Baseline (before hospital discharge), 3-Months Post-Surgery
Population: Number of participants who answered at least one followup anxiety survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Arm | Intervention
Number analyzed (Participants) | 11195 | 15227
score on a scale
  Baseline | 50.72 (9.20) | 51.85 (9.17)
  Month 1 | 51.93 (9.34) | 51.63 (9.59)
  Month 2 | 51.21 (9.54) | 51.75 (9.49)
  Month 3 | 47.19 (9.55) | 47.48 (9.62)

4. Primary Outcome: Use of Non-Pharmacological Pain Control Modalities
Description: Number of participants using Non-Pharmacological Pain Control Modalities
Time Frame: 3 Months Post-Surgery
Population: Patients who answered a questionnaire about their use of non-pharmacologic pain control modalities
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention
Number analyzed (Participants) | 958 | 25142
Participants
  Acupressure | 23 | 752
  Aromatherapy | 58 | 2549
  Cold or Heat | 721 | 16058
  Relaxed Breathing | 278 | 10709
  Guided Imagery | 23 | 1024
  Massage | 303 | 6848
  Meditation | 166 | 4254
  Muscle Relaxation | 183 | 5436
  Music | 184 | 7545
  Tai Chi | 7 | 257
  TENS | 58 | 1359
  Walking | 630 | 17886
  Yoga | 27 | 1237

5. Primary Outcome: Opioid Use
Description: Binary variables indicating presence or absence of opioid administration and prescription during the hospital encounter associated with the index surgery and during the post-discharge follow-up period.
Time Frame: 3-Months Post-Surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention
Number analyzed (Participants) | 25088 | 43054
Participants
  Any opioid administered in hospital associated with index surgery (excluding day of surgery) | 16158 | 26035
  Any opioid prescribed at discharge following index surgery | 19082 | 30414
  Any opioid prescription or administration associated with index surgical encounter | 22299 | 37639
  Any opioid administered inpatient during post-hospitalization follow-up period | 4972 | 7238
  Any opioid prescribed during post-hospitalization follow-up period | 7348 | 10422
  Any opioid prescription written during study period | 20173 | 31738
  Any opioid exposure (prescription or inpatient administration) during study period | 23034 | 38654

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for up to 3 Months Post-Surgery for all participants. Sites were monitored for the duration of the study (40 months)
Description: All deaths and adverse events were collected irrespective of attribution. No deaths or adverse events were causally associated with the NOHARM trial intervention.
Arm/Group | Control Arm | Intervention
All-Cause Mortality (participants affected / at risk) | 380/25088 | 608/43054
Serious Adverse Events (participants affected / at risk) | 25/25088 | 104/43054
Other Adverse Events (participants affected / at risk) | 2897/25088 | 4766/43054
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Arm (N=25088) | Intervention (N=43054)
Fall (General disorders) | 25 | 104 — Fall during index hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Arm (N=25088) | Intervention (N=43054)
Rash (Skin and subcutaneous tissue disorders) | 521 | 886 — Rash during study period
Muscle spasm (Musculoskeletal and connective tissue disorders) | 338 | 612 — Muscle spasm during study period
Failure to rescue (General disorders) | 2012 | 3234 — Failure to reduce pain: 3 or more consecutive severe pain scores (>= 7 on numeric rating scale out of 10)
Burn at electrode or hot pack site (Skin and subcutaneous tissue disorders) | 26 | 34 — Burn at electrode of hot pack site during study period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/71/NCT04570371/Prot_SAP_004.pdf